CLINICAL TRIAL: NCT04481477
Title: Impact on Patients of Nurses' Emotional Support Activities During Hospital Admission With a Diagnosis of COVID19
Brief Title: Results of Emotional Support Activities During Hospital Admission With a Diagnosis of COVID19
Acronym: WW2COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Montserrat Montaña, Principal Investigator, Clinical Research, Corporacion Parc Tauli
Other Study IDs: 2020664
Record Dates: First submitted 2020-07-21; First posted 2020-07-22 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Covid19
Keywords: Nursing care; Anxiety; Loneliness; Fear; COVID-19
MeSH Terms: conditions — COVID-19; Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients COVID-19: Patients over the age of 18 who were admitted with a diagnosis of COVID-19 to any CCSPT unit between March 13, 2020 and April 30, 2020 and were discharged with a recovery result
  Interventions: Other: Nursing care to reduce anxiety, fear and loneliness

INTERVENTIONS:
Other: Nursing care to reduce anxiety, fear and loneliness — Decreased anxiety Presence Emotional support Improved security Increasing coping capacity Presence Emotional support Facilitating visits

SUMMARY:
The aim of the study is to find out what care patients affected by anxiety, fear or loneliness have perceived and the perceived impact of this care. This knowledge will allow us to design measures aimed at improving nursing care of these aspects in the future.

DETAILED DESCRIPTION:
This is a cross-sectional descriptive study to be carried out at the Consorci Corporació Sanitària Parc Taulí (CCSPT). The results of this study will provide information on the care received by patients admitted to COVID 19 affected by anxiety, fear or loneliness, the perceived impact of this care and will enable measures to be implemented to improve nursing care in the future. 450 patients, randomly selected from the Hospital de Sabadell database, will be included. In the sample, we will ensure that the proportion of women and men is in line with the distribution of the population to enable the incorporation of the gender perspective in the analyses. The quantitative variables will be described by means of their mean and standard deviation. Qualitative variables will be described in absolute and relative frequencies. In order to evaluate the suitability of the intervention to the needs of the patient, a table of concordance will be constructed between the actions proposed by the panel of experts and the actions carried out as referred by the patient. The kappa concordance index will be calculated and the degree of concordance will be classified according to the Landis and Koch scale. As regards the effectiveness of the intervention, the patients who were treated correctly and those who were not will be identified, and the percentage of positive impacts according to Csq-8 between the two groups will be compared by means of the Chi-square test.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 who were admitted with a diagnosis of COVID-19 to any CCSPT unit between March 13, 2020 and April 30, 2020 and were discharged with a recovery result

Exclusion Criteria:

* Communication problems or inability to read and speak Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Residents in the CCSPT reference area
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2020-11-27 (Actual); Primary Completion 2021-04-15 (Estimated); Study Completion 2021-04-15 (Estimated)

PRIMARY OUTCOMES:
The adequacy of nursing care to the needs of the patient | 6 months after care
  kappa concordance rate between care provided and care needed

SECONDARY OUTCOMES:
Intervention effectiveness | 6 months after care
  comparison of the percentage of positive impacts according to Csq-8 between the two groups using the Chi-square test

CONTACTS AND LOCATIONS:
Overall Officials: Montserrat Montaña, PhD, Principal Investigator — Corporación Parc Taulí
Locations (1):
- CorporacionPT, Sabadell, Barcelona, Spain